CLINICAL TRIAL: NCT05743517
Title: Patient-Tailored Physical Activity Intervention Among Older Women With Gynecologic Cancers Undergoing Chemotherapy (Fit4Treatment)
Brief Title: Physical Activity Intervention Among Older Women With Gynecologic Cancers (Fit4Treatment)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Emma Barber, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00218257
Record Dates: First submitted 2023-01-31; First posted 2023-02-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Ovary Cancer; Endometrial Cancer; Uterine Cancer; Cervical Cancer; Cervix Cancer; Vulvar Cancer; Vaginal Cancer
Keywords: behavioral intervention; physical activity; cancer outcomes; chemotherapy; systemic therapy; quality of life
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The researchers will use a MOST full factorial study design to optimize the Fit4Treatment physical activity intervention by testing the core intervention of an activity tracker and commercially available app (Fitbit) in addition to four components which are expected to improve physical activity: 1) symptom-burden tailored goal setting app, 2) exercise partner, 3) oncology provider engagement, and 4) coaching calls. Patients will be randomized to 16 groups formed by all possible combinations of these four components in a full factorial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Symptom burden-tailored goal setting app (Experimental): The Fit4Treatment app is designed to encourage physical activity among older women with gynecologic cancer while they are undergoing cancer therapy. The app will contain the following features 1) education about safely increasing physical activity and steps; 2) tailored patient-specific push notifications to encourage physical activity 3) syncing of Fitbit steps and transmission of these data to study staff in real time; 4) daily, weekly and monthly step progress; and 5) goal setting that incorporates prior physical activity, patient desires, and daily symptom burden. The app will prompt patients to report their symptom burden on a scale of 1-5 each morning. Based on their symptom rating and the previous days step counts (measured directly by the Fitbit) patients will be provided with three different goal choices to select. Daily activity goals increase, decrease or stay the same depending on the previous day and the patient's own goals.
  Interventions: Behavioral: Fit4Treatment
- Exercise Partner (Experimental): Participants assigned to the exercise partner component will be encouraged to discuss their step progress with their selected partner who will in turn support the participant and encourage them to stay active.
  Interventions: Behavioral: Fit4Treatment
- Provider/oncologist engagement (Experimental): Participants assigned to the provider/oncologist engagement component will have their physical activity data recorded by the Fitbit shared with their oncology provider through the electronic medical record (EMR). For participants randomized to this condition, clinical staff will place an order into the EMR, allowing the patient to use the patient-facing portal MyChart to link their Fitbit to the health record. Prior to regularly scheduled clinic visits, the patient's oncology team will receive a message summarizing the participant's physical activity (average daily steps) for the prior three weeks.
  Interventions: Behavioral: Fit4Treatment
- Coaching (Experimental): Participants assigned to the coaching intervention will receive weekly coaching calls. The study team will call them at a previously specified and mutually agreed upon time once per week to review topics related to physical activity and cancer treatment. Coaching calls will have an educational component and cover topics such as reducing sedentary behavior, benefits of increased physical activity, managing cancer treatment symptoms, social support, stress management, etc. During these calls, the topics as well as strategies and recommendations will be discussed. Barriers and facilitators will be reflected on and planned for to increased self-efficacy. Participants will engage in direct problem solving with their coach. Discussing these topics will enhance outcome expectation and increase motivation.
  Interventions: Behavioral: Fit4Treatment

INTERVENTIONS:
Behavioral: Fit4Treatment — This study will test the core intervention of an activity tracker and commercially available app (Fitbit) in addition to four components which are expected to improve physical activity. The intervention will be delivered over 12 weeks with a 12 week follow up period.

SUMMARY:
The primary purpose of the study is to determine which of four components (symptom-burden tailored app, exercise partner, oncology provider engagement, coaching) added to a core intervention of a wearable activity tracker and commercially available app, will improve physical activity. The findings will generate meaningful knowledge about how to best increase physical activity in older gynecologic cancer patients receiving systemic cancer therapies to improve quality of life and cancer-specific survival.

DETAILED DESCRIPTION:
Gynecologic cancers include ovarian, uterine and cervical cancers and represent 102,000 cases of cancer in the United States every year; 60% occur in women greater than age 60. Older patients with gynecologic cancers have higher rates of advanced stage at presentation, more aggressive histology and more commonly require adjuvant treatment with systemic therapies such as chemotherapy, immunotherapy or targeted therapies. This chemotherapy, as well as underlying cancer, cause accelerated aging and toxicity, leaving women vulnerable to functional decline, increased frailty, decreased health related quality of life, and ultimately, less systemic therapy completion and inferior cancer survival.

Physical activity has been shown to improve functional health, improve quality of life, slow aging, and decrease rates of frailty. In fact, physical activity, and the multi-system health benefits that result, is the most recommended frailty intervention. Physical activity interventions in cancer survivors reduce sedentary time, decrease functional decline, and lower mortality. Studies specific to patients on active cancer treatment are less common, however, several randomized trials have found less decline in cardiorespiratory fitness, less chemotherapy toxicity, and fewer chemotherapy dose reductions. Although older adults with gynecologic cancer have a high likelihood of benefit from physical activity, challenges exist in accessing current interventions. Traditional in-person strenuous physical activity interventions with static goals may not be appropriate for older women undergoing chemotherapy, where symptom burden is high and varied, and healthcare visits frequent.

Remotely delivered mobile health (mHealth) technology-based physical activity interventions increase physical activity in diverse populations including those with metastatic cancer. Four evidence-based strategies to increase physical activity have demonstrated efficacy in cancer patients and older adults, including, 1) symptom burden tailored goal setting 2) exercise partners 3) oncology provider engagement and 4) coaching. This study will determine which components of a physical activity intervention (Fit4Treatment) meaningfully contribute to improving physical activity (steps) among older women with gynecologic cancer receiving systemic treatment such as chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female; > 60 years of age
* Diagnosis of endometrial/uterine, ovarian, cervical or vulvar/vaginal cancer
* Undergoing or planning to undergo any systemic treatment for a gynecologic malignancy (e.g., chemotherapy, immunotherapy, anti-angiogenic therapies, targeted therapies, etc.)
* Willing to try to identify an exercise partner to participate with them, if needed
* Fluent in English

Exclusion Criteria:

* Uncontrolled cardiovascular disease or other major contraindications to physical activity
* Active brain metastases
* Cognitive or functional limitations that preclude a patient's ability to participate in the physical activity intervention
* Pregnant women or prisoners

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity | 24 weeks
  The primary outcome of average steps per day over a 7 day period will be measured with Actigraph. Patients will wear an accelerometer for 7 days prior to study intervention, 7 days at the conclusion of the 12-week Fit4Treatment intervention, and 7 days at the conclusion of the 12 week follow up period.

SECONDARY OUTCOMES:
Change in Functional Performance | 24 weeks
  Patients will complete the short performance physical battery (SPPB). This is a well validated physical performance measure specifically in an older patient population and consists of balance testing, a 4-meter walk test and timed standing from a chair.
Change in Frailty | 24 weeks
  Frailty will be assessed using the Fried's phenotype method.
Change in Anxiety | 24 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) for anxiety will be measured at baseline, after the 12-week intervention, and after 24 weeks using Patient Reported Outcomes Measurement Information System Item Bank v1.0 - Emotional Distress - Anxiety - Short Form 7a, using a scale of 1-5, where 1 is the best outcome.
  PROMIS measures are validated, reliable measures of health states that can be completed with minimal patient burden and have been used in myriad studies of both older adults and cancer patients.
Change in Fatigue | 24 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) for fatigue will be measured at baseline, after the 12-week intervention, and after 24 weeks using Patient Reported Outcomes Measurement Information System Item Bank v1.0 - Fatigue - Short Form 7a, using a scale of 1-5, where 1 is the best outcome.
  PROMIS measures are validated, reliable measures of health states that can be completed with minimal patient burden and have been used in myriad studies of both older adults and cancer patients.
Change in Physical Function | 24 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) for physical function will be measured at baseline, after the 12-week intervention, and after 24 weeks using Patient Reported Outcomes Measurement Information System Item Bank v1.0 - Physical Function - Short Form 10a, using a scale of 1-5, where 1 is the best outcome.
  PROMIS measures are validated, reliable measures of health states that can be completed with minimal patient burden and have been used in myriad studies of both older adults and cancer patients.
Change in Pain Interference | 24 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) for pain will be measured at baseline, after the 12-week intervention, and after 24 weeks using Patient Reported Outcomes Measurement Information System Item Bank v1.0 - Pain Interference - Short Form 6a, using a scale of 1-5, where 1 is the best outcome.
  PROMIS measures are validated, reliable measures of health states that can be completed with minimal patient burden and have been used in myriad studies of both older adults and cancer patients.
Change in Sleep Disturbance | 24 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS) for sleep disturbance will be measured at baseline, after the 12-week intervention, and after 24 weeks using Patient Reported Outcomes Measurement Information System Item Bank v1.0 - Sleep Disturbance - Short Form 6a, using a scale of 1-5, where 1 or 5 is the best outcome, depending on the question.
  PROMIS measures are validated, reliable measures of health states that can be completed with minimal patient burden and have been used in myriad studies of both older adults and cancer patients.
Change in Global Quality of Life | 24 weeks
  Quality of Life will be measured at baseline, after the 12-week intervention, and after 24 weeks using the Global Quality of Life (QOL) scale of 1-5, where 5 is the best outcome.
Treatment Outcomes | 3 years
  Medical record review will be performed to examine treatment(s) administered and treatment delays.
Treatment Complications | 3 years
  Medical record review will be performed to monitor complications of systemic treatment.
Healthcare Utilization | 3 years
  Medical record review will be performed to monitor for hospitalizations, emergency room visits, and unscheduled clinic visits.
Survival Outcomes | 3 years
  Medical records will be reviewed for three years to monitor for cancer recurrence.
Adverse Events | 3 years
  The number of adverse events will be recorded and graded according to Common Terminology Criteria for Adverse Events, v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barber, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No